CLINICAL TRIAL: NCT00313326
Title: Comparative Study of Duration of Respiratory Weaning Between Adaptive Support Ventilation and Succession of Controlled Ventilation Then Spontaneous Ventilation for Patients After Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Dr Eric Schneider, CHU Clermont-Ferrand
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CHU63-005
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Ventilator Weaning
Keywords: Adaptive Support ventilation; Weaning

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: Adaptative Support Ventilation — Adaptive Support Ventilation (ASV) is a new protocol of weaning of the tracheal prosthesis after surgery which maintains a preset ventilation by an operator, and this whatever the activity of the patient

SUMMARY:
This is a comparative study of duration of respiratory weaning between adaptive support ventilation and succession of controlled ventilation then spontaneous ventilation for patients after surgery.

DETAILED DESCRIPTION:
General anaesthesia is marked by the passage of a stage of controlled ventilation where the patient does not carry out any respiratory work and the stage of spontaneous ventilation, which precedes extubation. Adaptive support ventilation (ASV) is a new protocol of weaning of the tracheal prosthesis after surgery which maintains a preset ventilation by an operator and the activity of the patient. At each breath, a microprocessor allows an optimization of volume and frequency by an adjustment of the inspiratory pressure and frequency. ASV was already validated for fast tracheal extubation after cardiac surgery. Our study proposes to compare the duration of intubation between this mode of weaning and with the traditional way (controlled ventilation then spontaneous ventilation) for faster surgery. The purpose of the study is to check the interest of ASV to limit the duration of intubation compared to the traditional protocol in this kind of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Surgery < 2 hours
* Anesthesia with thiopental, midazolam, sufentanil and suprane

Exclusion Criteria:

* Patients ASA III or IV (classification of American Sociéty of Anesthésiologist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2005-02; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Duration of weaning | duration

SECONDARY OUTCOMES:
Memorizing of weaning | memorizing

CONTACTS AND LOCATIONS:
Overall Officials: Eric Schneider, Doctor, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, France

REFERENCES:
- [Background] Petter AH, Chiolero RL, Cassina T, Chassot PG, Muller XM, Revelly JP. Automatic "respirator/weaning" with adaptive support ventilation: the effect on duration of endotracheal intubation and patient management. Anesth Analg. 2003 Dec;97(6):1743-1750. doi: 10.1213/01.ANE.0000086728.36285.BE. PMID 14633553
- [Background] Sulzer CF, Chiolero R, Chassot PG, Mueller XM, Revelly JP. Adaptive support ventilation for fast tracheal extubation after cardiac surgery: a randomized controlled study. Anesthesiology. 2001 Dec;95(6):1339-45. doi: 10.1097/00000542-200112000-00010. PMID 11748389